CLINICAL TRIAL: NCT01211301
Title: Randomized Controlled Trial of the Medifast 5 & 1 Plan
Brief Title: Medifast 5 & 1 Plan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Medifast, Inc. (Industry)
Responsible Party: Principal Investigator, David Allison, Phd, Prof/Assoc Dean, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F100625001
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Obesity; Body Weight; Weight Loss; Overweight; Nutrition Disorders
Keywords: obesity; overweight; weight loss; randomized controlled trial; Medifast
MeSH Terms: conditions — Obesity; Body Weight; Weight Loss; Overweight; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Food-based, Reduced Energy Diet Plan (Active Comparator)
  Interventions: Behavioral: Food-based, Reduced Energy Diet Plan
- Medifast 5 & 1 Plan (Experimental)
  Interventions: Other: Medifast 5 & 1 Plan

INTERVENTIONS:
Behavioral: Food-based, Reduced Energy Diet Plan — Control participants will be provided with a 1000-kcal/d meal plan based on regular foods selected and procured by participants. Food lists, sample menus, and portion size references will be provided.
  Arms: Food-based, Reduced Energy Diet Plan
Other: Medifast 5 & 1 Plan — Participants randomized to the Medifast group will enroll online in the Medifast 5 & 1 Plan. This plan consists of 5 portion-controlled, nutritionally-balanced Medifast Meals plus one Lean & Green Meal each day. Medifast Meals come in individual packets that are mixed with water and microwaved or refrigerated, and are available in a wide variety of foods and flavors. There are >70 Medifast Meal choices, and Medifast Meals may be used interchangeably, so any five Medifast Meals can be chosen for the 5 & 1 Plan. The Medifast 5 & 1 Plan provides approximately 800 to 1,000 kcal/d. The Lean & Green Meal consists of a lean meat plus salad and/or vegetables selected by the participant. Intervention participants will have online access to Medifast dietitians, Medifast trainers, a Medifast message board, and a Medifast chat room, allowing them to interact with others on the Medifast 5 & 1 Plan.
  Arms: Medifast 5 & 1 Plan

SUMMARY:
The purpose of this study is to compare the effectiveness of the Medifast 5 & 1 Plan to a food-based, reduced-energy diet plan. The study will be conducted over 52 weeks, including a 26-week weight-loss phase and a 26-week weight-maintenance phase. 120 participants will be enrolled, with 60 randomized to the Medifast 5 & 1 Plan and 60 randomized to food-based, reduced-energy diet plan. Multiple measures will be performed at baseline, 26 weeks, and 52 weeks, including anthropometry, body composition, blood pressure, blood assays, and appetite sensations.

ELIGIBILITY:
Inclusion Criteria:

* BMI 35-50 kg/m2
* Interested in weight loss
* Computer with internet access
* Any race or ethnicity
* Fasting glucose <126 mg/dL at screening

Exclusion Criteria:

* Participation in any weight-reduction program, weight-loss diet, or other special diet within the previous 3 months.
* Weight loss or gain of >5% body weight in past 6 months for any reason except post-partum weight loss.
* Currently taking any medication that suppresses or stimulates appetite.
* History of prior surgical procedure for weight control or liposuction.
* Current smoker or quit smoking less than 6 months prior.
* Any major disease, including:

  * Active cancer or cancer requiring treatment in the past 2 years (except nonmelanoma skin cancer).
  * Active or chronic infections, including self-reported HIV positivity and active tuberculosis.
  * Active cardiovascular disease or event including hospitalization or therapeutic procedures for treatment of heart disease (e.g., coronary artery bypass, percutaneous transluminal coronary angioplasty) in the past 6 months; New York Heart Association Functional Class >2 with respect to congestive heart failure; stroke or transient ischemic attack in the past 6 months.
  * Uncontrolled hypertension: systolic blood pressure >160 mm Hg or diastolic blood pressure >95 mm Hg on treatment.
  * Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
  * Active kidney disease.
  * Lung disease: chronic obstructive airway disease requiring use of oxygen.
  * Diagnosed diabetes (type 1 or 2), fasting hyperglycemia (blood glucose >126 mg/dL), or use of any anti-diabetic medications.
* Uncompensated or uncontrolled psychiatric disease (such as schizophrenia and bipolar disorder) that, in opinion of the investigators, would impede conduct of the trial or completion of procedures.
* A score on the Brief Symptom Inventory (BSI) (Derogatis & Melisaratos, 1983) that exceeds the 90th percentile.
* History of or current eating disorders, or an Eating Attitudes Test (EAT 40) score >30.
* Active food allergies, particularly to wheat, gluten, soy or nuts.
* Conditions or behaviors likely to effect the conduct of the trial: unable or unwilling to give informed consent; unable to communicate with the pertinent clinic staff; another household member is a participant or staff member in the trial; unwilling to accept treatment assignment by randomization; current or anticipated participation in another intervention research project that would interfere with the intervention offered in the trial; likely to move away from participating clinics before trial completed; unable to walk 0.25 mile in 10 minutes.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage is stable.
* No regular source of health care.
* Any active use of illegal or illicit drugs or history of illegal or illicit drug utilization within past year
* Excessive alcohol intake, either acute or chronic defined as any one of the following: 1) average consumption of 3 or more alcohol containing beverages daily; 2) consumption of 7 or more alcoholic beverages within a 24-hr period in the past 12 months; or 3) other evidence available to clinic staff.
* Willing to limit alcohol intake to zero
* Pregnancy and childbearing: currently pregnant or less than 3 months post partum; currently nursing or within 6 weeks of having completed nursing; pregnancy anticipated during study; unwilling to report possible or confirmed pregnancies promptly during the course of the trial; unwilling to take adequate contraceptive measures if potentially fertile.
* Any other conditions which, in opinion of the investigators, would adversely affect the conduct of the trial.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2012-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Body weight | 26 and 52 weeks

SECONDARY OUTCOMES:
Waist circumference | 26 and 52 weeks
Body composition as measured by bioelectrical impedence (BIA) | 26 and 52 weeks
Body mass index | 26 and 52 weeks
Low-density lipoprotein cholesterol (LDL) | 26 and 52 weeks
High-density lipoprotein cholesterol (HDL) | 26 and 52 weeks
Triglycerides | 26 and 52 weeks
Glucose | 26 and 52 weeks
Liver function tests | 26 and 52 weeks
High-sensitivity C-reactive protein (hs-CRP) | 26 and 52 weeks
Lipid hydroperoxides | 26 and 52 weeks
Blood pressure | 26 and 52 weeks
Appetite/satiety measures | 26 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David B. Allison, PhD., Principal Investigator — University of Alabama at Birmingham; James M. Shikany, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Division of Preventive Medicine, Birmingham, Alabama, United States

REFERENCES:
- [Result] Shikany JM, Thomas AS, Beasley TM, Lewis CE, Allison DB. Randomized controlled trial of the Medifast 5 & 1 Plan for weight loss. Int J Obes (Lond). 2013 Dec;37(12):1571-8. doi: 10.1038/ijo.2013.43. Epub 2013 Apr 9. PMID 23567927